CLINICAL TRIAL: NCT02394080
Title: CE Marking Study of the IlluminOss Photodynamic Bone Stabilization System for the Treatment of Humerus Fractures
Brief Title: Safety and Efficacy Study of the Treatment of Humerus Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IlluminOss Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-03-EUHUM-01; NCT02524314 (obsolete NCT alias)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Acute Humerus Fractures

ARMS (1):
- Photodynamic Bone Stabilization System (PBSS) (Experimental): The PBSS is comprised of an inflatable, thin walled polyethylene terephthalate (PET; Dacron™) balloon mounted on an insertion catheter. This balloon catheter system is designed to deliver the monomer cement to the fracture site via the medullary canal of the bone.
  Interventions: Device: Photodynamic Bone Stabilization System

INTERVENTIONS:
Device: Photodynamic Bone Stabilization System — Treatment of acute humerus fractures

SUMMARY:
The purpose of this study is to collect safety and performance data on the use of the Photodynamic Bone Stabilization System (PBSS) when used to provide stabilization and alignment for the treatment of acute humerus fractures.

ELIGIBILITY:
Fracture-Specific Inclusion Criteria

1. Radiograph-confirmed diagnosis of acute, single isolated fracture of the humerus. AO classification 11A2, 11A3 and 11B1, 11B2 and 12A1, 12A2, 12A3 and 12B1, 12B2.
2. Fracture is closed, Gustilo Type I or II.

   General Inclusion Criteria
3. Skeletally mature men and women, 50 years of age or older at time of index injury.
4. a) Female patients of child bearing potential agree to use double barrier method of contraception b) Female patients of non-child bearing potential must meet one of the following criteria:

   * Postmenopausal for at least 1 year, or
   * Documented oophorectomy or hysterectomy, or
   * Surgically sterile
5. Willing and able to understand and sign the informed consent.

Fracture-Specific Exclusion Criteria

1. Index treatment is greater than 28 days post fracture
2. Open fractures with severe contamination.
3. Extremely comminuted fractures where insufficient holding power of the balloon on the intramedullary canal is probable.
4. Marked bone loss or bone resorption patients, who due to a prior delayed union or non-union of the bones or other illnesses, may not be able to have their fracture adequately reduced prior to placement of the IlluminOss-device. This could leave bone void spaces that would preclude the device from maintaining alignment of the fractured bone.
5. Previous fracture of affected limb.

   General Exclusion Criteria
6. Pregnant or lactating.
7. Active or incompletely treated infections that could involve the site where the device will be implanted.
8. Distant foci of infections that may spread to the implant site
9. Uncooperative patients or patients, who are incapable of following directions (for example as a consequence of a neurological or psychiatric disorder).
10. Concomitant metabolic disorders that may impair bone formation.
11. Osteomalacia.
12. Allergic to implant materials or dental glue.
13. Vascular insufficiency, muscular atrophy, or neuro-muscular disease.
14. Polytrauma patients (multiple injuries resulting from a high-impact event, eg- a motor vehicle accident).
15. Life expectancy less than one year due to concurrent illness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Normal radiographic fracture healing | 180 days
  Two of four cortices or two of four views demonstrating bridging on standard radiographs

SECONDARY OUTCOMES:
Assessment of the incidence of adverse events | 180 and 360 days
Assessment of the procedure- and device-related complication rate | 180 and 360 days
Evaluation of complete radiographic healing | 180 and 360 days
  Three of four cortices or three of four views demonstrating bridging, with dissolution of the majority (greater than or equal to 75% on orthogonal views) of fracture lines
Evaluation of normal radiographic healing | 360 days
  Two of four cortices or two of four views demonstrating bridging on standard radiographs
Assessment of no pain at palpation status | 180 and 360 days
  Clinical assessment
Assessment of return to pre-fracture mobility status | 180 and 360 days
  Clinical assessment
Comparison of pain visual analog score (VAS) from baseline to all follow up intervals | 180 and 360 days
Comparison of Disability of the Arm, Shoulder and Hand score from baseline to all follow up intervals | 180 and 360 days
Comparison of Constant shoulder score from baseline to all follow up intervals | 180 and 360 days
Assessment of range of motion | 180 and 360 days
  Clinical assessment
Assessment of disability status | 180 and 360 days
  Per Investigator assessment
Assessment of return to work status | 180 and 360 days

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amphia Hospital, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - University Hospital Maastricht, Maastricht